CLINICAL TRIAL: NCT00718237
Title: A Phase III Randomized, Placebo-controlled Clinical Trial to Study the Efficacy and Safety of V260 in Healthy Infants in Japan
Brief Title: Phase III Placebo-controlled Study of V260 (RotaTeq™) in Japanese Healthy Infants (V260-029)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V260-029; 2008_014
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2010-07-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Rotavirus; Gastroenteritis
Keywords: Gastroenteritis; Rotavirus
MeSH Terms: conditions — Gastroenteritis | interventions — Rotavirus Vaccines; RotaTeq

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): RotaTeq™
  Interventions: Biological: Rotavirus Vaccine, Live, Oral, Pentavalent (V260, RotaTeq™)
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Comparator: Placebo (unspecified)

INTERVENTIONS:
Biological: Rotavirus Vaccine, Live, Oral, Pentavalent (V260, RotaTeq™) — Rotateq orally administered 3 times
  Other Names: RotaTeq™; V260
  Arms: 1
Biological: Comparator: Comparator: Placebo (unspecified) — Placebo orally administered 3 times
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate whether V260 is effective and well tolerated in Japanese healthy infants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Japanese Infants, 6 Weeks Through 12 Weeks Of Age

Exclusion Criteria:

* History Of Known Prior Rotavirus Gastroenteritis
* Subjects Who Are Concurrently Participating In Or Are Anticipated To Participate In Other Studies Of Investigational Products At Any Time During The Study Period

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 762 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Iwata S, Nakata S, Ukae S, Koizumi Y, Morita Y, Kuroki H, Tanaka Y, Shizuya T, Schodel F, Brown ML, Lawrence J. Efficacy and safety of pentavalent rotavirus vaccine in Japan: a randomized, double-blind, placebo-controlled, multicenter trial. Hum Vaccin Immunother. 2013 Aug;9(8):1626-33. doi: 10.4161/hv.24846. Epub 2013 May 31. PMID 23732903

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 32 sites in Japan from 2008 to 2009.
Pre-assignment Details: Excluded from the trial before assignment to groups were subjects with: history of congenital abdominal
  disorders, intussusception, or abdominal surgery; history of known prior rotavirus disease, chronic diarrhea,
  or failure to thrive; immune impairment or resides in a household with an individual with an immune impairment.
Groups:
- RotaTeq™: Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with 14 days of safety follow-up after each vaccination, and follow-up for acute gastrointestinal episodes (AGEs) until the end of the study.
- Placebo: Three doses of placebo matching RotaTeq™ administered 28 to 70 days apart, with 14 days of follow-up after each vaccination, and follow-up for AGEs until the end of the study.
Period: Overall Study
Arm/Group | RotaTeq™ | Placebo
Started | 381 (Subjects who passed all entry criteria and who were randomized into the study) | 381 (Subjects who passed all entry criteria and who were randomized into the study)
Vaccinated at Visit 1 | 380 | 381
Vaccinated at Visit 2 | 373 | 374
Vaccinated at Visit 3 | 371 | 369
Completed | 368 (Subjects who continued follow-up until the last visit, regardless of number of vaccinations received) | 366 (Subjects who continued follow-up until the last visit, regardless of number of vaccinations received)
Not Completed | 13 | 15
Not completed — Adverse Event | 1 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 9 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RotaTeq™ | Placebo | Total
Number analyzed (Participants) | 381 | 381 | 762
Age, Continuous [Mean (Standard Deviation); unit: Weeks] | 7.6 (1.7) | 7.5 (1.6) | 7.5 (1.6)
Age, Customized [Number; unit: participants]
  6 to 12 Weeks of age | 381 | 381 | 762
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173 | 182 | 355
  Male | 208 | 199 | 407

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Moderate to Severe Rotavirus Gastroenteritis Caused by Rotavirus Serotypes G1, G2, G3, G4 and G-serotypes Associated With Serotype P1A
Description: Moderate to severe cases of rotavirus gastroenteritis caused by G1, G2, G3, G4 or G-serotypes associated with serotype P1A occurring at least 14 days postdose 3 in the per-protocol population using per-protocol case definition. Severity score was calculated based on frequency and duration of diarrhea, vomiting, elevated temperature, and behavioral changes. Score of >8 and <=16 was considered moderate, and >16 was considered severe.
Time Frame: At least 14 days following the 3rd vaccination
Population: Per Protocol Population; number randomized is different from number analyzed due to some data excluded from the analysis (e.g., protocol violators, unevaluable due to detection of wild-type rotavirus in stool prior to 14 days Postdose 3, incomplete clinical and/or laboratory results, or stool samples collected out of day range).
Measure: Number; unit: Number of participants
Groups:
- RotaTeq™: Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with 14 days of follow-up after each vaccination, and follow-up for AGEs until the end of the study.
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 354 | 356
Number of participants | 5 [47.4 to 94.1] | 25
Statistical Analysis 1: Comparison: RotaTeq™; Test type: Superiority or Other; p < 0.001, Exact Conditional Test — Hypothesis: Efficacy >0%. Based on p< 1/(1+k); p = proportion of participants with outcome in vaccine group relative to total number of subjects with outcome; k = ratio of follow-up time; placebo/vaccine. Based on conditional binomial approach; Exact Conditional Test based on Binomial Distribution; Vaccine Efficacy (1-Relative Risk [RR]) = 80.2, 95% CI 2-sided [47.4 to 94.1] — Efficacy = 1-RR, expressed as a percentage; the RR is the incidence in the vaccine group / the incidence in the placebo group, adjusted for the ratio of the follow-up period in each group

2. Primary Outcome: Number of Participants With Rotavirus Gastroenteritis of Any Severity Caused by Rotavirus Serotypes G1, G2, G3, G4 and G-serotypes Associated With Serotype P1A
Description: Any severity cases of rotavirus gastroenteritis caused by G1, G2, G3, G4 or G-serotypes associated with serotype P1A occurring at least 14 days postdose 3 in the per-protocol population using per-protocol case definition
Time Frame: At least 14 days following the 3rd vaccination
Population: as for outcome 1
Measure: Number; unit: Number of participants
Groups:
- RotaTeq™: Three doses of RotaTeq™ (Rotavirus vaccine, live, oral, pentavalent) administered 28 to 70 days apart, with 14 days of follow-up after each vaccination, and follow-up for acute gastrointestinal episodes (AGEs) until the end of the study.
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 355 | 356
Number of participants | 7 [39.9 to 90.6] | 27
Statistical Analysis 1: Comparison: RotaTeq™; Test type: Superiority or Other; p < 0.001, Exact Conditional Test — [p-value comment as in outcome 1, analysis 1]; Exact Conditional Test based on Binomial Distribution; Vaccine Efficacy (1-Relative Risk [RR]) = 74.5, 95% CI 2-sided [39.9 to 90.6] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Participants With Severe Rotavirus Gastroenteritis Caused by Rotavirus Serotypes G1, G2, G3, G4 and G-serotypes Associated With Serotype P1A
Description: Severe cases of rotavirus gastroenteritis caused by G1, G2, G3, G4 or G-serotypes associated with serotype P1A occurring at least 14 days postdose 3 in the per-protocol population using per-protocol case definition. Severity score was calculated based on frequency and duration of diarrhea, vomiting, elevated temperature, and behavioral changes. Score of >8 and <=16 was considered moderate, and >16 was considered severe.
Time Frame: At least 14 days following the 3rd vaccination
Population: Per Protocol Population; number randomized is different from number analyzed due to some data excluded from the analysis (e.g., protocol violators, unevaluable due to detection of wild-type rotavirus in stool antigen prior to 14 days Postdose 3, incomplete clinical and/or laboratory results, or stool samples collected out of day range).
Measure: Number; unit: Number of participants
Arm/Group | RotaTeq™ | Placebo
Number analyzed (Participants) | 354 | 355
Number of participants | 0 [55.4 to 100.0] | 10
Statistical Analysis 1: Comparison: RotaTeq™; Test type: Superiority or Other; p < 0.001, Exact Conditional Test — [p-value comment as in outcome 1, analysis 1]; Exact Conditional Test based on Binomial Distribution; Vaccine Efficacy (1-Relative Risk [RR]) = 100.0, 95% CI 2-sided [55.4 to 100.0] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 14-day period following each vaccination. Any death, Vaccine related SAE and Intussusception were collected during the study period.
Description: Parents/guardians were asked to record AEs on a standardized Vaccine Report Card (VRC) during 14 days after each vaccination. Solicited AEs included diarrhea and vomiting. Temperature was also measured daily for 7 days after each vaccination.
  The number of patients listed "At Risk" is the number of patients who received study treatment.
Arm/Group | RotaTeq™ | Placebo
Serious Adverse Events (participants affected / at risk) | 7/380 | 9/381
Other Adverse Events (participants affected / at risk) | 179/380 | 175/381
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ (N=380) | Placebo (N=381)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1
Congenital absence of bile ducts (Congenital, familial and genetic disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Meningitis coxsackie viral (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Infantile spasms (Nervous system disorders) | 0 | 1
Psychomotor retardation (Psychiatric disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RotaTeq™ (N=380) | Placebo (N=381)
Conjunctivitis (Eye disorders) | 7 | 3
Constipation (Gastrointestinal disorders) | 11 | 7
Diarrhoea (Gastrointestinal disorders) | 46 | 47
Infantile spitting up (Gastrointestinal disorders) | 6 | 2
Vomiting (Gastrointestinal disorders) | 31 | 29
Pyrexia (General disorders) | 29 | 31
Bronchitis (Infections and infestations) | 7 | 8
Gastroenteritis (Infections and infestations) | 27 | 14
Nasopharyngitis (Infections and infestations) | 37 | 37
Respiratory syncytial virus infection (Infections and infestations) | 4 | 2
Rhinitis (Infections and infestations) | 0 | 8
Upper respiratory tract infection (Infections and infestations) | 4 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 27 | 16
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 9 | 6
Eczema (Skin and subcutaneous tissue disorders) | 14 | 12
Eczema infantile (Skin and subcutaneous tissue disorders) | 7 | 10
Rash (Skin and subcutaneous tissue disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.